CLINICAL TRIAL: NCT02077881
Title: A Phase I/II Study of Indoximod in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Study of IDO Inhibitor in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG2104
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Metastatic Pancreatic Cancer
Keywords: metastatic; metastasis; Pancreatic; Pancreas; Cancer; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms; Adenocarcinoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel; Gemcitabine; 1-methyltryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indoximod and Gemcitabine + Nab-paclitaxel (Experimental): Phase 1 portion:
  Participants to receive indoximod (600mg, 100mg, or 1200mg according to their assigned dose cohort) PO BID for 28 days concurrently with IV Nab-paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 weekly for 3 weeks with one week rest. Each cycle is 28 days. Patients will continue until they experience disease progression or significant toxicity.
  Phase 2 portion:
  Once a RP2D is determined, treatment will commence with oral indoximod concurrent with the first backbone chemotherapy cycle.Patients will receive gemcitabine plus nab-paclitaxel on a standard 4 week cycle schedule. Oral indoximod will continue throughout.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Indoximod

INTERVENTIONS:
Drug: Nab-Paclitaxel — Nab-Paclitaxel 125 mg/m^2 given intravenously over 30-40 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest. Patients will continue until they experience disease progression or significant toxicity.
  Other Names: Abraxane; Paclitaxel
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 given intravenously over 30 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest. Patients will continue until they experience disease progression or significant toxicity.
  Other Names: Gemzar
Drug: Indoximod — Indoximod will be administered in escalating doses. Initial dosing will be 600 mg BID by mouth with escalation planned to 1200 mg BID by mouth
  Indoximod in the form of 200 mg capsules will be given (3, 5, and 6 capsules depending on the escalated dose). Indoximod should be taken with water by mouth one hour before breakfast and one hour prior to dinner. The medication should be taken twice daily for 28 days each cycle. Patients will continue until they experience disease progression or toxicity.
  Other Names: 1-methyl-D-tryptophan; D-1MT

SUMMARY:
This phase I/II trial is designed to efficiently identify the regimen limiting toxicity (RLT) and recommended phase 2 dose (RP2D) for the combination of the immunotherapeutic agent indoximod when administered in combination with standard of care chemotherapy gemcitabine plus nab-paclitaxel in subjects with metastatic adenocarcinoma of the pancreas. All subjects will receive the same standard gemcitabine plus nab-paclitaxel regimen, plus indoximod in doses increasing from 600 mg twice daily to, potentially, 1200 mg twice daily.

DETAILED DESCRIPTION:
This is a Phase I/II trial designed to evaluate the combination of the immunotherapeutic agent indoximod and the standard of care chemotherapy gemcitabine plus nab-paclitaxel in subjects with metastatic adenocarcinoma of the pancreas. The phase 1 portion is designed to identify the regimen-limiting toxicity (RLT) and recommended phase 2 dose (RP2D) for the combination. The phase 2 portion of the study will evaluate the potential efficacy of this combination. All subjects will receive the standard 28-day gemcitabine plus nab-paclitaxel regimen. Twice daily oral indoximod will be administered concurrently in continuous 28 day cycles.

In the phase 1 portion, dose escalation of indoximod will begin at 600 mg twice a day and potentially escalate to 1200 mg twice a day. There will be no intra-subject dose escalation. Regimen-limiting toxicity will be considered as those toxicities related to indoximod that significantly limit the administration of the backbone chemotherapy gemcitabine plus nab-paclitaxel. The period for determination of dose-limiting toxicities will be the initial 28 days of treatment. The recommended phase 2 dose will include an assessment of toxicities that occur at later time points.

Once a RP2D is determined, the phase 2 portion of the study will be initiated. In both phase 1 and phase 2, every 2 cycles subjects will have repeat imaging to assess response. Corollary biomarkers will be assessed at the same interval as will PET-CT after the 1st 8 week cycle. Up to 18 patients will be enrolled in the phase 1 portion of the study and 80 patients will be enrolled in the phase 2 portion.

ELIGIBILITY:
Inclusion Criteria:

* Patient has definitive histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. Patients with islet cell or neuroendocrine neoplasms are excluded.
* Initial diagnosis of metastatic disease must have occurred ≤8 weeks prior to entry in the study.
* Patient has one or more metastatic tumors measurable per RECIST 1.1 by CT scan ≤4 weeks prior to entry into the study
* Male or non-pregnant and non-lactating female, and ≥18 years of age.
* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease.
* Prior treatment with gemcitabine and/or nab-paclitaxel in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Patients cannot have received any other immunomodulatory therapies (including vaccines) as treatment for this or any other cancer.
* Patient has a Karnofsky performance status (KPS) ≥ 70.
* Patients should be asymptomatic for jaundice prior to Day 1.

Exclusion Criteria:

* Patients may not be receiving (or received prior to enrollment) any other investigational agents for metastatic disease.
* Patient has known brain metastases,
* Patient has only locally advanced disease.
* Lymph node only metastases even if considered M1 disease by official staging criteria.
* History of malignancy in the last 3 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 3 years.
* Patients with any active autoimmune disease
* Patient has undergone major surgery, other than diagnostic surgery (ie, surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Phase 2 Dosing | 10 months
  Phase 1 component:
  To determine recommended phase 2 dose of indoximod when administered with a standard of care chemotherapy backbone consisting of gemcitabine plus nab-paclitaxel.
Regimen Limiting Toxicity | 10 months
  Phase 1 component:
  To identify the regimen limiting toxicity (RLT) for the combination of the immunotherapeutic agent indoximod when administered in combination with standard of care chemotherapy gemcitabine plus nab-paclitaxel in subjects with metastatic adenocarcinoma of the pancreas.
  RLT will be considered as only grade 3 and 4 toxicities that are attributable to the test agent and result in the delay of the administration of the backbone chemotherapy, gemcitabine plus nab-paclitaxel.
Overall Survival | 22 months
  Phase 2 component:
  To evaluate efficacy as determined by overall survival (OS) in patients with metastatic adenocarcinoma of the pancreas.

SECONDARY OUTCOMES:
Biomarker Response | 22 months
  A secondary objective is to examine biomarker responses of gemcitabine and nab-paclitaxel with indoximod through the evaluation of serum for biomarkers of IDO activity (kynurenine and tryptophan), before and after initiation of therapy through specimen collection at protocol specified timepoints.
Response Rate | 22 months
  To determine the response rate of the combination indoximod with gemcitabine plus nab-paclitaxel. Imaging assessments to be performed at protocol-specified time points and evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
Time to Progression of Disease | 22 months
  To determine the time to progression with the combination indoximod with gemcitabine plus nab-paclitaxel. Progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Augusta University, Augusta, Georgia
  - University of Kentucy, Lexington, Kentucky
  - Washington University in St. Louis, St Louis, Missouri
  - The Vally Hospital, Paramus, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Health Systems, Greenville, South Carolina
  - Gibbs Cancer Center and Research Institute, Spartanburg, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Huntsman Cancer Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Derived] Beatty GL, Delman D, Yu J, Liu M, Li JH, Zhang L, Lee JW, Chang RB, Bahary N, Kennedy EP, Wang-Gillam A, Rossi GR, Garrido-Laguna I. Treatment Response in First-Line Metastatic Pancreatic Ductal Adenocarcinoma Is Stratified By a Composite Index of Tumor Proliferation and CD8 T-Cell Infiltration. Clin Cancer Res. 2023 Sep 1;29(17):3514-3525. doi: 10.1158/1078-0432.CCR-23-0535. PMID 37534996